CLINICAL TRIAL: NCT04934540
Title: The Global En Bloc Resection of Bladder Tumour Registry
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Jeremy Yuen Chun TEOH, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: CRE 2020.369
Record Dates: First submitted 2020-11-11; First posted 2021-06-22 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Bladder Cancer
Keywords: En bloc resection of bladder tumour
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing ERBT: Patients who are diagnosed with bladder tumors and planning for ERBT.
  Interventions: Procedure: En bloc resection of bladder tumour

INTERVENTIONS:
Procedure: En bloc resection of bladder tumour — En bloc resection of bladder tumour (ERBT) is a novel surgical technique in which the bladder tumour is resected in one piece

SUMMARY:
The study aims to collect data on ERBT globally in order to clarify its role in the management of bladder cancer over a 5-year observation period.

DETAILED DESCRIPTION:
Bladder cancer is a prevalent disease globally, and it is the 9th most commonly diagnosed cancer in men worldwide. It has a standardized incidence rate of 9.0 per 100,000 person-years for men and 2.2 per 100,000 person-years for women. This disease represents a significant burden to the healthcare system.

Bladder cancer is classified into non-muscle-invasive bladder cancer (NMIBC) and muscle-invasive bladder cancer (MIBC) according to its depth of invasion. Conceptually, NMIBC is amenable to complete resection by transurethral resection of bladder tumour (TURBT) alone, while MIBC requires more aggressive treatment in the form of radical cystectomy. The gold standard in local staging is by histology, and this can be achieved by TURBT. However, conventional TURBT creates charred tissue chips in a piecemeal manner which may hinder pathologists' judgment of the tumour base clearance. Second-look TURBT has been shown to detect residual disease in 33-55% of the patients, and upstaging of disease in 4-45% of the patients following the first TURBT; it has also been shown to improve recurrence-free survival in patients with T1 non-muscle-invasive bladder cancer. In addition, tumour fragmentation and reimplantation may lead to early disease recurrence. All these highlighted the limitations of the conventional TURBT procedure.

Transurethral en bloc resection of bladder tumour (ERBT) represents a novel surgical technique in which the bladder tumour is resected in one piece. Theoretically, ERBT may prevent recurrence by minimizing the risk of tumour reimplantation and ensuring complete resection based on proper histological assessment. Although ERBT has been practised in many centres worldwide, there is a lack of high quality evidence in proving its superiority over conventional TURBT. Also, the optimal indications, best energy modality, the need for routine tumour base biopsy, intravesical chemotherapy, second-look TURBT and the optimal follow-up protocol remain uncertain for this technique. Therefore, there is a need for a well-planned prospective multi-centre study to evaluate the role of ERBT in the management of bladder cancer.

Investigators propose to conduct a prospective, multi-centre, registry study to expedite understanding of ERBT and to establish its role in management of bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >=18 years old with informed consent
* Presence of bladder tumour undergoing transurethral ERBT

Exclusion Criteria:

* Presence or previous history of upper tract urothelial carcinoma
* Presence of other active malignancy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed with bladder tumors upon flexible cystoscopy and planning for ERBT
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The complete tumour resection rate | One weeks after the surgery
  Complete tumour resection refers to successful ERBT with negative circumferential and deep resection margins.
Recurrence-free survival for NMIBC | Every 3 months for the first two years, and then every 6 months for the next three years.
  Recurrence-free survival for patients with non-muscle-invasive bladder cancer

SECONDARY OUTCOMES:
Proper staging rate for NMIBC | Seven weeks after the operation
  The proper staging rate for NMIBC is defined as the absence of any upstaging of the T-stage upon second-look TURBT or radical surgery, in patients who have NMIBC upon the first ERBT. Second look transurethral resection surgery or radical surgery are expected to perform within six weeks after the first operation and one more week is allowed for histological assessment of the second operative specimen.
Proper staging rate for MIBC | Seven weeks after the operation
  The proper staging for MIBC is defined as the detection of MIBC upon the first En bloc resection, in all patients who have a definitive histological diagnosis of MIBC upon second-look TURBT or radical surgery. Second look transurethral resection surgery or radical surgery are expected to perform within six weeks after the first operation and one more week is allowed for histological assessment of the second operative specimen
Complete tumour resection rate for MIBC | Seven weeks after the operation
  The complete tumour resection rate for MIBC is defined as the absence of any malignancy upon second-look TURBT or radical surgery, in patients who have MIBC upon the first ERBT. Second look transurethral resection surgery or radical surgery are expected to perform within six weeks after the first operation and one more week is allowed for histological assessment of the second operative specimen
Successful ERBT rate | Immediately post-operative
  Technical success rate of en bloc resection
Negative circumferential resection margin rate | One week after the operation
  Rate of negative circumferential resection margin of the en bloc resection pathological specimen
Negative deep resection margin rate | One week after the operation
  Rate of negative deep resection margin of the en bloc resection pathological specimen
Detrusor muscle sampling rate | One week after the operation
  Rate of presence of detrusor muscle in the en bloc resection pathological specimen
Occurrence of obturator reflex | Intra-operative
  Number of participants with obturator reflex encountered by the operating surgeon during the en bloc resection operation
Operative time | Immediately post-operative
  Duration of operation
Rate of mitomycin C instillation | Immediately post-operative
  One day after the surgery
Duration of bladder irrigation | Three days after the operation
  Duration of bladder irrigation. Patients undergoing transurethral resection surgery have an average hospital stay of three days. Bladder irrigation is always stopped before the patient is discharged
Hospital stay | Three days after the operation
  Patients undergoing transurethral resection surgery have an average hospital stay of three days.
30-day complications | Thirty days after the operation
  The 30-day complications will be graded according to the Clavien-Dindo classification
Progression-free survival | Every 3 months for the first two years, and then every 6 months for the next three years.
  Progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy YC TEOH, FRCS(Ed) MBBS, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - North District Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Grimm MO, Steinhoff C, Simon X, Spiegelhalder P, Ackermann R, Vogeli TA. Effect of routine repeat transurethral resection for superficial bladder cancer: a long-term observational study. J Urol. 2003 Aug;170(2 Pt 1):433-7. doi: 10.1097/01.ju.0000070437.14275.e0. PMID 12853793
- [Background] Divrik RT, Sahin AF, Yildirim U, Altok M, Zorlu F. Impact of routine second transurethral resection on the long-term outcome of patients with newly diagnosed pT1 urothelial carcinoma with respect to recurrence, progression rate, and disease-specific survival: a prospective randomised clinical trial. Eur Urol. 2010 Aug;58(2):185-90. doi: 10.1016/j.eururo.2010.03.007. Epub 2010 Mar 19. PMID 20303646
- [Background] Jahnson S, Wiklund F, Duchek M, Mestad O, Rintala E, Hellsten S, Malmstrom PU. Results of second-look resection after primary resection of T1 tumour of the urinary bladder. Scand J Urol Nephrol. 2005;39(3):206-10. doi: 10.1080/00365590510007793-1. PMID 16127800
- [Background] Lazica DA, Roth S, Brandt AS, Bottcher S, Mathers MJ, Ubrig B. Second transurethral resection after Ta high-grade bladder tumor: a 4.5-year period at a single university center. Urol Int. 2014;92(2):131-5. doi: 10.1159/000353089. Epub 2013 Aug 23. PMID 23988813
- [Background] Vasdev N, Dominguez-Escrig J, Paez E, Johnson MI, Durkan GC, Thorpe AC. The impact of early re-resection in patients with pT1 high-grade non-muscle invasive bladder cancer. Ecancermedicalscience. 2012;6:269. doi: 10.3332/ecancer.2012.269. Epub 2012 Sep 18. PMID 22988482
- [Background] Simon R, Eltze E, Schafer KL, Burger H, Semjonow A, Hertle L, Dockhorn-Dworniczak B, Terpe HJ, Bocker W. Cytogenetic analysis of multifocal bladder cancer supports a monoclonal origin and intraepithelial spread of tumor cells. Cancer Res. 2001 Jan 1;61(1):355-62. PMID 11196186
- [Background] Babjuk M, Bohle A, Burger M, Capoun O, Cohen D, Comperat EM, Hernandez V, Kaasinen E, Palou J, Roupret M, van Rhijn BWG, Shariat SF, Soukup V, Sylvester RJ, Zigeuner R. EAU Guidelines on Non-Muscle-invasive Urothelial Carcinoma of the Bladder: Update 2016. Eur Urol. 2017 Mar;71(3):447-461. doi: 10.1016/j.eururo.2016.05.041. Epub 2016 Jun 17. PMID 27324428
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542